CLINICAL TRIAL: NCT01826331
Title: Incentives for Participation Versus Outcomes for Population Cessation of Smoking
Brief Title: Incentives for Participation Versus Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator died
Sponsor: University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: DA034041
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (No Intervention): Participants will be incentivized for assessments only
- Incentives for Participation (Experimental): Participants will be incentivized for each assessment and for each smoking cessation session they complete
  Interventions: Behavioral: Incentives for Participation
- Incentives for Cessation (Experimental): Participants will be incentivized for each assessment and biochemically confirmed abstinence at 12 and 24 months
  Interventions: Behavioral: Incentives for Cessation

INTERVENTIONS:
Behavioral: Incentives for Participation — Participants will receive three smoking cessation programs
  Arms: Incentives for Participation
Behavioral: Incentives for Cessation — Participants will have access to a smoking cessation program
  Arms: Incentives for Cessation

SUMMARY:
One of the most important debates in the field of disease prevention is whether financial incentives should be contingent on participation in evidence-based programs for smoking cessation or on actual outcomes, like prolonged abstinence. This study can fill a major knowledge gap in this debate, which is the lack of any population trial that compared the impacts of outcomes- and participation-based incentives in a population of smokers. This research can help policy makers and health service providers choose the incentives approach that provides the most effectiveness, cost-effectiveness and cost-savings for entire populations of smokers.

DETAILED DESCRIPTION:
This population-based randomized clinical trial is designed to compare long-term abstinence rates in three groups of smokers: 1. Those incentivized for participation in an evidence-based treatment designed for smokers at each stage of change; 2. Those incentivized for biologically validated prolonged abstinence at 6 and 12 months who could also choose to participate in the TTM (Transtheoretical Model)-tailored intervention; and 3. An assessment only control condition.

The Specific Aims are:

1. To assess whether the treatment group incentivized for participation outperforms the control group at 12, 24 and 36 months as hypothesized;
2. To assess whether the treatment group incentivized for prolonged abstinence at 6 and 12 months outperforms the control group at each follow-up as hypothesized;
3. To assess whether the treatment group incentivized for participation outperforms the treatment group incentivized for outcomes at 36 months as hypothesized.
4. To compare the cost-effectiveness of each treatment in a population of mostly unmotivated smokers;

The Secondary Aims are:

1. To assess the long-term treatment trajectories of each treatment compared to controls with hypothesized increasing trajectory in the participation contingent incentives and decreasing trajectory in the outcome contingent incentives.
2. To identify mediators of long-term outcomes in each treatment, such as amount of treatment participation, income, severity of smoking, stage of change, self-efficacy, perceived health and intrinsic and extrinsic motivation to quit.
3. To compare cost-savings of each treatment by modeling all additional costs of smoking for employers and smokers.

ELIGIBILITY:
Inclusion Criteria:

* smoker

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James O Prochaska, Ph.D., Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States